CLINICAL TRIAL: NCT00740259
Title: Is Flunarizine a Cheap, Well-Tolerated and Long-Acting Atypical Antipsychotic? A Randomized Double-Blind Flexible-Dose Clinical Trial Versus Haloperidol for the Treatment of Schizophrenia
Brief Title: Efficacy and Tolerability of Flunarizine for the Treatment of Schizophrenia: Comparison With Haloperidol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ambulatório de Bipolaridade (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Diogo Rizzato Lara, Ambulatório de Bipolaridade
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Flunarizine for schizophrenia; 02T-264 (SMRI)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia
Keywords: flunarizine; schizophrenia; antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Flunarizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Flunarizine — For 1 week, 40 mg/day. From week 2 to 3, 20 mg/day. Form week 4 onwards, dosage increment or reduction of 10mg/day was allowed according to efficacy and tolerability.

SUMMARY:
Flunarizine is a calcium channel blocker traditionally used for the treatment of vertigo and migraine. It also has the mechanism of action associated with antipsychotic activity (D2 receptor blockade), but has never been tested as such. The investigators hypothesis is that flunarizine can be an atypical antipsychotic.

DETAILED DESCRIPTION:
The main advantage of flunarizine over other D2 receptor blockers is its long half-life, so that it may be administered weekly or may delay relapse if medication is interrupted.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV schizophrenic or schizoaffective patients between 18 and 55 years old with a PANSS score above 45.

Exclusion Criteria:

* Clinical disease
* Pregnancy
* Drug dependence (except for nicotine) in the past month and history of being refractory to at least 2 antipsychotics taken appropriately.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2004-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Bisol LW, Brunstein MG, Ottoni GL, Ramos FL, Borba DL, Daltio CS, de Oliveira RV, Paz GE, de Souza SE, Bressan RA, Lara DR. Is flunarizine a long-acting oral atypical antipsychotic? A randomized clinical trial versus haloperidol for the treatment of schizophrenia. J Clin Psychiatry. 2008 Oct;69(10):1572-9. doi: 10.4088/jcp.v69n1007. Epub 2008 Sep 1. PMID 19192440